CLINICAL TRIAL: NCT03489941
Title: A Single-Center Evaluation of the Relative Efficacy of EM-100 Compared to Zaditor® (Ketotifen Fumarate Ophthalmic Solution 0.035%) and Vehicle in the Treatment of Ocular Itching Associated With Allergic Conjunctivitis as Induced by the Conjunctival Allergen Challenge Model (Ora-CAC®)
Brief Title: A Single-Center Evaluation of the Relative Efficacy of EM-100 Compared to Zaditor® (Ketotifen Fumarate Ophthalmic Solution 0.035%) and Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-100-0011
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2021-04

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — ketotifen fumarate ophthalmic solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- EM-100 (Experimental): One drop of EM-100 in either the right or left eye once on Day 1.
  Interventions: Drug: EM-100
- Zaditor® (Experimental): One drop of Zaditor® in either the right or left eye once on Day 1.
  Interventions: Drug: Zaditor®
- Vehicle (Experimental): One drop of Vehicle in either the right or left eye once on Day 1.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: EM-100 — Subjects will receive one drop in one eye only based on the randomization list, one time over the course of the trial.
  Arms: EM-100
Drug: Zaditor® — Subjects will receive one drop in one eye only based on the randomization list, one time over the course of the trial.
  Arms: Zaditor®
Drug: Vehicle — Subjects will receive one drop in one eye only based on the randomization list, one time over the course of the trial.
  Arms: Vehicle

SUMMARY:
A Single-Center study to demonstrate the non-inferiority of EM-100 to Zaditor® in the treatment of ocular itching.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years old
* have a positive history of allergic conjunctivitis and positive skin test reaction to allergens
* be willing to avoid disallowed medications for the appropriate washout period and throughout the trial
* be willing to avoid contact lens use
* be willing to have a pregnancy test
* must be able to read an eye chart from 10 feet away

Exclusion Criteria:

* must not have any allergies to the study medications
* must not have any ocular or non ocular condition that investigator feels will interfere with study parameters
* must not have used an investigational drug or device in the past 30 days or currently be enrolled in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Total Eye Care, PA, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 65 participants enrolled (130 eyes). 38 participants received EM-100 in one eye and Zaditor in the other eye. 13 participants received EM-100 in one eye and vehicle in the other eye. 14 participants received Zaditor in one eye and vehicle in the other eye. Thus, of 65 participants, 51 received EM-100 in one of their eyes, 52 received Zaditor in one of their eyes, and 27 received vehicle in one of their eyes. Each participant received 2 of the 3 study treatments, one in each eye.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | EM-100 | Zaditor® | Vehicle
Started | 51; 51 eyes | 52; 52 eyes | 27; 27 eyes
Completed | 51; 51 eyes | 52; 52 eyes | 27; 27 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: The 65 enrolled participants had one of the three study treatments instilled in each eye (each subject had 2 of the 3 different treatments, one in each eye). Demographic data were not collected by treatment or by eye.
Arm/Group | Overall Participants
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 36
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Iris color [Count of Participants; unit: Participants]
  Black | 1
  Blue | 8
  Brown | 46
  Hazel | 6
  Green | 4

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching scores were self-assessed by the participant using a 5-point scale with 0.5 unit increments, wherein 0 = None (normal, no itching), 1.0 = Intermittent tickle sensation involving more than just the corner of the eye, 2.0 = Mild continuous itch without desire to rub, 3.0 = Severe itch with desire to rub, and 4.0 = Incapacitating itch with irresistible urge to rub.
Time Frame: 3, 5 and 7 minutes post-Conjunctival Allergen Challenge (CAC) on Day 1
Population: The 65 enrolled participants had one of the three study treatments instilled in each eye (each subject had 2 different treatments, one in each eye).
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | EM-100 | Zaditor® | Vehicle
Number analyzed (Participants) | 51 | 52 | 27
Number analyzed (eyes) | 51 | 52 | 27
score on a scale
  3 minutes post CAC | 0.81 (0.787) | 0.79 (0.750) | 1.98 (0.935)
  5 minutes post CAC | 1.09 (1.047) | 1.04 (0.989) | 2.17 (1.00)
  7 minutes post CAC | 1.17 (1.103) | 1.04 (1.047) | 2.22 (1.032)

2. Secondary Outcome: Conjunctival Redness
Description: The investigator assessed conjunctival redness scores using a 5-point scale with 0.5 unit increments, wherein 0 = None (normal, no dilated blood vessels), 1 = Mild (slightly dilated blood vessels: pink color; can be quadrantal), 2 = Moderate (more apparent dilation, with redder color, involving majority of the vessel bed), 3 = Severe (numerous and obvious dilated blood vessels, with deep red color and no color, or less red with chemosis), and 4 = Extremely Severe (large, numerous, dilated blood vessels characterized by unusually severe deep red color regardless of chemosis and involving the entire vessel bed).
Time Frame: 7, 15 and 20 minutes post-Conjunctival Allergen Challenge (CAC) on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EM-100 | Zaditor® | Vehicle
Number analyzed (Participants) | 51 | 52 | 27
score on a scale
  7 minutes post-CAC | 2.13 (0.824) | 2.14 (0.743) | 2.72 (0.725)
  15 minutes post-CAC | 2.25 (0.783) | 2.29 (0.737) | 2.61 (0.847)
  20 minutes post-CAC | 2.16 (0.857) | 2.24 (0.704) | 2.46 (0.784)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Overall Participants: The 65 enrolled participants had one of the three study treatments instilled in each eye (each subject had 2 of the 3 different treatments, one in each eye).
Arm/Group | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03489941/Prot_SAP_001.pdf